CLINICAL TRIAL: NCT00951405
Title: An Exploratory Multi-Centre, Multi-National, Randomised, Double Blinded, Parallel Arm Trial Evaluating Safety, Pharmacokinetics and Dose-finding of Prophylactic Administration of Long Acting rFVIIa (LA-rFVIIa) in Haemophilia A or B Patients With Inhibitors
Brief Title: Safety and Efficacy of 3 Different Doses of Long Acting Factor VII in Haemophilia A or B Patients With Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NN7128-1907; 2008-006424-54 (EudraCT Number); JapicCTI-090860 (Registry Identifier: JAPIC); U1111-1111-8584 (Other: WHO)
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental)
  Interventions: Drug: activated recombinant human factor VII, long acting
- B (Experimental)
  Interventions: Drug: activated recombinant human factor VII, long acting
- C (Experimental)
  Interventions: Drug: activated recombinant human factor VII, long acting

INTERVENTIONS:
Drug: activated recombinant human factor VII, long acting — After an observation period of 3 months, every 2nd day intravenous (i.v.) injection with 25 microgrammes/kg activated recombinant human factor VII, long acting, for 3 months
  Other Names: NN7128; LA-rFVIIa
  Arms: A
Drug: activated recombinant human factor VII, long acting — After an observation period of 3 months, every 2nd day intravenous (i.v.) injection with 100 microgrammes/kg activated recombinant human factor VII, long acting, for 3 months
  Other Names: NN7128; LA-rFVIIa
  Arms: B
Drug: activated recombinant human factor VII, long acting — After an observation period of 3 months, every 2nd day intravenous (i.v.) injection with 200 microgrammes/kg activated recombinant human factor VII, long acting, for 3 months
  Other Names: NN7128; LA-rFVIIa
  Arms: C

SUMMARY:
This trial is conducted in Asia, Europe, Japan and North America. The aim of this clinical trial is to investigate the safety and the efficacy of a prophylactic treatment option with long acting coagulation factor VII (LA-rFVIIa) for haemophilia patients with inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Male haemophilia A or B patients with inhibitors
* Willing to undergo a bleeding preventive regimen of 3 months' duration and a total trial length of approximately 8 months
* Historical or ongoing high titre inhibitor (more than or equal to 5 BU) based on either medical records, laboratory report reviews, patient and/or care provider interviews
* At least 2 bleeding episodes requiring bypassing haemostatic-drug-based treatment within the last month or 12 bleeding episodes within the last 6 months prior to observation period
* Body weight between 30 and 100 kg (both inclusive)

Exclusion Criteria:

* Body Mass Index (BMI) above 30 kg/m2
* Immune tolerance induction therapy within the last month prior to entering observation phase period
* Known active pseudo tumours
* Platelet count less than 50,000 platelets/microL (based on local laboratory value at screening visit)
* Congenital or acquired coagulation disorders other than haemophilia A or B
* Surgery within one month prior to the observation period. Catheter, stents and dental extractions do not count as surgeries, i.e. they will not exclude the patient. Port insertion is classified as surgery
* Scheduled major and/or orthopaedic surgery, during the trial period until Follow up visit. Catheter, stents and dental extractions do not count as surgeries and will not exclude the patient. Port insertion is classified as surgery
* Advanced atherosclerotic disease (i.e. known history of ischemic heart disease, or ischemic stroke)
* Any clinical signs or known history of thromboembolic events incl. known deep vein thrombosis (DVT)
* Known or clinically suspected allergy to activated recombinant human factor VII (NovoSeven®/NovoSeven RT®/Niastase®)
* Prothrombin Time (PT) prolongation (30% above normal limits, or more than 5 seconds compared to control or International Normalised Range (INR) more than 1.7 as defined by local laboratory ranges at screening visit
* Severe liver disease (ALAT more than 4 times of the upper limit of normal reference range) (as defined by local laboratory ranges) within a year of enrolment or at the screening
* Clinical signs of renal dysfunction (dialysis) and/or creatinine levels more than or equal to 20% above upper normal limit (according to local laboratory range at the screening visit)
* Dosing of any investigational drug within the last 30 days prior to the present trial
* Any disease or condition which, according to the investigator's judgement, could imply a potential hazard to the subject, interfere with the trial participation or trial outcome
* HIV positive patients who either have low CD4+ lymphocyte count ( 200/microL or less based on medical records within 6 months or laboratory screening at screening visit), or who are HCV-PCR positive (based on medical records), or who both have low CD4+ lymphocyte count (200/microL or less) and are HCV-PCR positive. If HCV-PCR testing is not locally available, a HIV positive patient who is HCV antibody positive cannot be included
* Need to use other PEGylated pharmaceutical drug during the trial period

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2011-03-29 (Actual); Study Completion 2011-03-29 (Actual)

PRIMARY OUTCOMES:
Thrombogenecity | at all scheduled visits (1 - 9)
Immunogenecity: Neutralising Antibody Development | at all scheduled visits (1 - 9)

SECONDARY OUTCOMES:
AUC(0-48h) and AUC: Area under the FVIIa activity-time profile in the given time period, which is a measure of total blood exposure | at visit 2 and visit 7 until 48 hours after trial product administration
Annualized bleeding rates | During observation period; from visit 1 until visit 2 and treatment period; from visit 2 until visit 7. In total a period of 6 to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (24):
- United States (7):
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
- Novo Nordisk Investigational Site, Rio de Janeiro, Brazil
- France (2):
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Paris
- Japan (4):
  - Novo Nordisk Investigational Site, Kashihara-shi, Nara
  - Novo Nordisk Investigational Site, Kitakyusyu, Fukuoka
  - Novo Nordisk Investigational Site, Nishinomiya-shi
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Belgrade, Serbia and Montenegro
- Novo Nordisk Investigational Site, Belgrade, Serbia
- South Africa (2):
  - Novo Nordisk Investigational Site, Parktown Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
- Novo Nordisk Investigational Site, Malmo, Sweden
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Istanbul
- United Kingdom (2):
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Oxford

REFERENCES:
- [Derived] Ljung R, Karim FA, Saxena K, Suzuki T, Arkhammar P, Rosholm A, Giangrande P; Pioneer1 Investigators. 40K glycoPEGylated, recombinant FVIIa: 3-month, double-blind, randomized trial of safety, pharmacokinetics and preliminary efficacy in hemophilia patients with inhibitors. J Thromb Haemost. 2013 Jul;11(7):1260-8. doi: 10.1111/jth.12237. PMID 23578227
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com